CLINICAL TRIAL: NCT03156699
Title: The Incidence, Effect and Persistence of Fragmented-QRS, in Patients Presenting With ST-Elevation Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: The Royal Wolverhampton Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2017CAR93
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: ST Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- STEMI patients treated with primary PCI: Database analysis only

SUMMARY:
This study will assess the incidence, effect and persistence of F-QRS (Fragmented-QRS) in STEMI (ST-elevation Myocardial Infarction) patients post-PCI (percutaneous coronary intervention). The aim is to add to the existing research field surrounding F-QRS. It is hypothesised that patients with F-QRS present on the surface ECG, following PCI, will have incurred a higher degree of damage. As a result, it is hypothesised that these patients will have reduced LV (left-ventricular) systolic function, increased incidence of regional wall motion abnormalities (RWMAs), and increased troponin levels on admission. This study will additionally look for correlations between F-QRS and culprit vessels. To our knowledge there is minimal research regarding this.

DETAILED DESCRIPTION:
This is a Physiological - Retrospective data collection from STEMI patients. Data from 100 STEMI patients treated with primary PCI will be extracted.

Data will be collected from presentation / initial admission, 6-week post-MI (Myocardial Infarction) clinic and 6 month post-MI clinic from the hospital system at New Cross Hospital. Data from admission includes; 12-lead ECG, echo reports and blood test results. Additionally, the 12-lead ECGs undertaken at 6-week and 6-months will be assessed for the presence of F-QRS.

ELIGIBILITY:
Inclusion Criteria:

* Look back to data at least 12 months old in order to ensure 6-week and 6-month follow up data is available. The inclusion criteria will be patients that presented with STEMI and were treated with primary PCI.

Exclusion Criteria:

* From the cath lab reports and clinical letters exclusions apply to patients that did not present with STEMI. In addition, patients that were not treated with primary PCI, or patients that deceased prior, during or post procedure (during hospitalization).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 100 STEMI patients treated with primary PCI.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
F-QRS measurements | Over 6 months
  recorded from ECG

SECONDARY OUTCOMES:
Left ventricular ejection fraction (LVEF) | Over 6 months
  recorded from ECG
T-Troponin tests | Over 6 months
  T-Troponin tests as cardiac biomarker of myocardial damage

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Kelly, Principal Investigator — The Royal Wolverhampton NHS Trust
Locations (1):
- New Cross Hospital, Wolverhampton, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No IPD will be available to other researchers